CLINICAL TRIAL: NCT01063660
Title: Clinical Phase II Trial to Evaluate the Safety and Efficacy of Treosulfan Based Conditioning Prior to Allogeneic Haematopoietic Stem Cell Transplantation in Patients With Acute Myeloid Leukaemia
Brief Title: Treosulfan Based Conditioning Acute Myeloid Leukaemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Prof. Dr. Mathias Freund, University of Rostock
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC-FludT.7/AML
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Acute Myeloid Leukaemia
Keywords: Treosulfan; Fludarabine; ATG; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treosulfan (Experimental): Patients with acute myeloid leukaemia (AML) according to WHO classification (> 20% myeloblasts in peripheral blood or bone marrow at initial diagnosis) with < 5% myeloblasts in the bone marrow, indicated for allogeneic transplantation
  Interventions: Drug: Treosulfan

INTERVENTIONS:
Drug: Treosulfan — 14 g/m²/d day -6 to -4
  Other Names: Ovastat

SUMMARY:
This is a multicenter, multinational, non-randomized, non-controlled open-label phase II trial to evaluate the safety and efficacy of treosulfan in a combination regimen with fludarabine as conditioning therapy prior to allogeneic stem cell transplantation (SCT) in patients with AML.

The aim is to demonstrate a clinical benefit compared with historical data on intravenous busulfan (BusulfexTM, BusilvexTM), the only drug so far registered in the indication conditioning before allogeneic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myeloid leukaemia (AML) according to WHO classification (> 20% myeloblasts in peripheral blood or bone marrow at initial diagnosis) with < 5% myeloblast in the bone marrow, indicated for allogeneic transplantation
* Availability of an HLA-identical sibling donor (MRD) or HLA-identical unrelated donor (MUD) HLA-identity defined by the following markers: A, B, DRB1, DQB1.
* Target graft size (unmanipulated)
* bone marrow: 2 - 10 x 106 CD34+ cells/kg BW recipient or > 2 x 108 nucleated cells/kg BW recipient or
* peripheral blood: 4 - 10 x 106 CD34+ cells/kg BW recipient
* Age > 18 and < 60 years
* Karnofsky Index > 80 %
* Adequate contraception in female patients of child-bearing potential
* Written informed consent

Exclusion Criteria:

* Therapy related secondary AML
* AML with t(8;21)(q22;q22) in CR1
* Acute promyelocytic leukaemia with t(15;17)(q22;q12) in CR1
* Secondary malignancies
* Previous allogeneic transplantation
* Severe concomitant illnesses / medical conditions (e.g. impaired respiratory and/or cardiac function)
* Known and manifested malignant involvement of the CNS
* Active infectious disease
* HIV- positivity or active hepatitis infection
* Impaired liver function (Bilirubin > upper normal limit; Transaminases > 3.0 x upper normal limit)
* Impaired renal function (Creatinine-clearance < 60 ml/min; Serum Creatinine > 1.5 x upper normal limit).
* Pleural effusion or ascites > 1.0 L
* Pregnancy or lactation
* Known hypersensitivity to treosulfan and/or fludarabine
* Participation in another experimental drug trial within 4 weeks before day -6
* Non-co-operative behaviour or non-compliance
* Psychiatric diseases or conditions that might impair the ability to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2004-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Efficacy - Evaluation of engraftment. Safety - Evaluation of the incidence of the following CTC grade 3 and 4 adverse events between day -6 and day +28 - hyperbilirubinemia and mucositis / stomatitis - veno-occlusive disease - seizures | 3.5 years

SECONDARY OUTCOMES:
Efficacy - Evaluation of disease free survival (DFS) - Evaluation of overall survival (OS) - Evaluation of relapse incidence (RI) - Donor chimerism on day +28, +56 and +100. Safety - Evaluation of NRM on days +28 and +100 | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Freund, MD, Principal Investigator — University of Rostock
Locations (1):
- University of Rostock, Rostock, Germany

REFERENCES:
- [Derived] Casper J, Holowiecki J, Trenschel R, Wandt H, Schaefer-Eckart K, Ruutu T, Volin L, Einsele H, Stuhler G, Uharek L, Blau I, Bornhaeuser M, Zander AR, Larsson K, Markiewicz M, Giebel S, Kruzel T, Mylius HA, Baumgart J, Pichlmeier U, Freund M, Beelen DW. Allogeneic hematopoietic SCT in patients with AML following treosulfan/fludarabine conditioning. Bone Marrow Transplant. 2012 Sep;47(9):1171-7. doi: 10.1038/bmt.2011.242. Epub 2011 Dec 12. PMID 22158386